CLINICAL TRIAL: NCT06694337
Title: Study to Investigate the Potential Pharmacological Effect of Oral Palmitoylethanolamide (PEA) Therapy in the Management of Low Back Pain (Neuropathic Pain): A Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Trial
Brief Title: Study to Investigate the Potential Pharmacological Effect of Oral Palmitoylethanolamide (PEA) Therapy in the Management of Low Back Pain (Neuropathic Pain)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LUMHS/REC/-531/25.11.2024
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — palmidrol; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 300 mg Palmitoylethanolamide (PEA) group (Experimental): Participants will receive 2 × 300 mg oral PEA Phytosome® tablets daily for one week, and a single tablet from week-7 to week-8, as add-on to the standard of care.
  Interventions: Dietary Supplement: 300 mg Palmitoylethanolamide (PEA) Phytosome®
- 450 mg Palmitoylethanolamide (PEA) group (Experimental): Participants will receive 1 × 450 mg oral PEA Phytosome® tablet, and 1 placebo tablet daily for 8-weeks as add-on to the standard of care.
  Interventions: Dietary Supplement: 450 mg Palmitoylethanolamide (PEA) Phytosome®; Other: Control group
- Control group (Placebo Comparator): Participants will receive 2 × placebo tablets daily for 8-weeks as add-on to the standard of care.
  Interventions: Other: Control group

INTERVENTIONS:
Dietary Supplement: 300 mg Palmitoylethanolamide (PEA) Phytosome® — Oral supplement intake
  Arms: 300 mg Palmitoylethanolamide (PEA) group
Dietary Supplement: 450 mg Palmitoylethanolamide (PEA) Phytosome® — Oral supplement intake
  Arms: 450 mg Palmitoylethanolamide (PEA) group
Other: Control group — Placebo
  Arms: 450 mg Palmitoylethanolamide (PEA) group; Control group

SUMMARY:
This clinical trial aims to evaluate the potential therapeutic effects of oral supplemental Palmitoylethanolamide (PEA) Phytosome® in managing neuropathic low back pain. The study will involve adult participants diagnosed with neuropathic pain according to established criteria. Eligible participants will be randomized into three groups to receive either PEA Phytosome® supplementation as two different doses or a placebo for a specified period. Data collection will include demographic information, baseline pain intensity, quality of life assessments, and functional outcomes. The primary endpoint will be the reduction in pain intensity, while secondary endpoints will include improvements in quality of life and functional capacity. Safety and tolerability of the supplement will also be assessed. This trial seeks to provide robust clinical evidence of the potential pharmacological effect of PEA's Phytosome® as a potential adjunctive treatment for neuropathic low back pain.

DETAILED DESCRIPTION:
Neuropathic low back pain arises from nerve damage or dysfunction, leading to chronic pain characterized by burning, tingling, or shooting sensations. This condition significantly impacts quality of life and is often refractory to conventional treatments. Palmitoylethanolamide (PEA) is an endogenous lipid mediator known for its anti-inflammatory, analgesic, and neuroprotective properties. PEA exerts its effects by modulating the endocannabinoid system and reducing the activation of mast cells and glial cells, which play a crucial role in chronic pain mechanisms. Its potential as a therapeutic agent for neuropathic pain has been demonstrated in preclinical and clinical studies, making it a promising candidate for managing neuropathic low back pain.

In the present randomized, double-blind, placebo-controlled, parallel-group clinical trial, the investigators aim to evaluate the therapeutic effect of a novel bioavailable oral formulation of PEA's Phytosome® in the management of neuropathic low back pain in healthy adult population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, both Male or female aged ≥ 18 years and ≤ 80 years;
* Diagnosed with neuropathic lower back pain for at least 3 months, as confirmed by clinical evaluation and DN4 (neuropathic pain 4 questions) screening questionnaire with score ≥4.
* Pain intensity score ≥ 5 measured by NRS (Numerical Rating Scale) score, over the past week.
* Willingness to adhere to study protocol, including visits, assessments, and self-reporting of symptoms.
* Ability to provide informed consent and comply with study requirements.

Exclusion Criteria:

* Known intolerance or allergy to any component of the tested nutraceuticals
* Presence of acute systemic disease
* Presence of significant organic pathology
* Current or past history of alcohol or drug abuse
* History of malignancy within the past 5 years
* Any significant concomitant disease or clinical condition that could compromise participant safety or interfere with study completion
* Women of childbearing potential not using reliable contraceptive methods
* Pregnancy or breastfeeding
* Severe psychiatric disorders (e.g., major depression, schizophrenia) that could affect pain perception or adherence.
* Inability to adhere to the study requirements due to lifestyle, transportation, or cognitive impairment.
* Use of other cannabinoid-based therapies, investigational drugs, or concurrent participation in another clinical trial.
* Dependence on opioid analgesics or recent opioid use that may interfere with pain assessment.
* Current use of other supplements with potential anti-inflammatory or analgesic effects, including Omega-3 Fatty Acids, Turmeric/Curcumin, Glucosamine and Chondroitin, Boswellia Serrata, Methylsulfonylmethane.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Supplement effect on neuropathic low back symptoms pain as experienced by the patients | 8 weeks
  Change in The Douleur Neuropathique 4 (DN4) questionnaire score, a 10-item, clinician-administered tool used to identify neuropathic pain. A score of 4 or more out of 10 is the cut-off for defining the presence of neuropathic pain.
Supplement effect on intensity of neuropathic low back pain | 8 weeks
  Change in neuropathic pain intensity measured by the Numerical Rating Scale (NRS) score, with 0 representing no pain and 10 representing the worst pain.

SECONDARY OUTCOMES:
Supplement effect on patients degree of disability | 8 weeks
  Change in degree of disability due to neuropathic back pain assessed by Oswestry Disability Index (ODI) questionnaire. A score of 0-20% indicates minimal disability, 21-40% moderate disability, 41-60% severe disability, 61-80% crippled, and 81-100% bedridden or completely disabled.
Supplement effect on patients quality of life | 8 weeks
  Short Form Health Survey 12 (SF-12) questionnaire score. The SF-12 questionnaire assesses quality of life through 12 items, producing two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Higher scores on both components indicate better physical and mental health, respectively.
Supplement effect on patients sleep quality | 8 weeks
  Change in patients sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI) score. A score of 5 or higher suggests clinically significant sleep disturbances.
Change in the number of times the rescue Non-steroidal anti-inflammatory drugs (NSAIDs) needed per week | 8 weeks
  Change in the weekly NSAIDs doses intake

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Reading Hospital, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keppel Hesselink JM, Kopsky DJ. Palmitoylethanolamide, a neutraceutical, in nerve compression syndromes: efficacy and safety in sciatic pain and carpal tunnel syndrome. J Pain Res. 2015 Oct 23;8:729-34. doi: 10.2147/JPR.S93106. eCollection 2015. PMID 26604814
- [Background] Clayton P, Hill M, Bogoda N, Subah S, Venkatesh R. Palmitoylethanolamide: A Natural Compound for Health Management. Int J Mol Sci. 2021 May 18;22(10):5305. doi: 10.3390/ijms22105305. PMID 34069940